CLINICAL TRIAL: NCT04926194
Title: Decidual Stromal Cells (DSC) in Treatment of Steroid-Refractory Graft-vs-host Disease in a Recipient of Matched Related Donor Allogeneic Hematopoietic Cell Transplant for Myelodysplastic Syndrome/Myeloproliferative Neoplasm
Brief Title: Decidual Stromal Cells to Treat Graft-vs-Host Disease After Stem Cell Transplant for Myelodysplastic Syndrome/Myeloproliferative Neoplasm
Acronym: DSC-SR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC-SR
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasm; Steroid Refractory GVHD; Allogeneic Hematopoietic Cell Transplant
MeSH Terms: conditions — Myelodysplastic-Myeloproliferative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with MDS/MPN (Experimental): DSCs will be given 1 × 10^6 cells per kilogram of participant's body weight intravenously, administered once per week up to a maximum of six weeks depending on the clinical response.
  Interventions: Biological: Decidual stromal cells (DSC)

INTERVENTIONS:
Biological: Decidual stromal cells (DSC) — DSCs are isolated from donated human placenta and have been shown to have anti-inflammatory effects.

SUMMARY:
This is a single participant study of decidual stromal cells (DSC) for the treatment of steroid refractory graft-versus-host disease (GVHD) in a patient with myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN).

ELIGIBILITY:
A single participant with myelodysplastic syndrome/myeloproliferative neoplasm located at Princess Margaret Cancer Centre who experienced steroid-refractory graft-vs-host disease after receiving an allogeneic hematopoietic cell transplant and have no standard treatment options available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Eastern Cooperative Oncology Group Performance Status Score | 6 weeks
Karnofsky Performance Score | 6 weeks
Graft-Versus-Host Disease Severity | 6 weeks
  By grade
Aspartate Transaminase levels | 6 weeks
Alanine aminotransferase levels | 6 weeks
Alkaline phosphatase levels | 6 weeks
Bilirubin levels | 6 weeks
C-reactive protein levels | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pasic, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No